CLINICAL TRIAL: NCT03238677
Title: Treating Childhood Apraxia of Speech: Role of Biofeedback & Practice Distribution
Brief Title: Treating Childhood Apraxia of Speech
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Jonathan Preston, Associate Professor, Syracuse University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 17-177; R15DC016426 (NIH)
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Childhood Apraxia of Speech
Keywords: speech sound disorder
MeSH Terms: conditions — Apraxias; Speech Sound Disorder | interventions — Biofeedback, Psychology

STUDY DESIGN:
Intervention Model Description: 2 x 2 design Scheduling: Mass-->Distributed vs. Distributed only Visual feedback: Sequenced Ultrasound Biofeedback vs. No biofeedback
Who Masked: Outcomes Assessor
Masking Description: Individuals who conduct the phonetic transcriptions that will be used for the primary outcome data will be blinded as to whether the recordings were collected before or after treatment, and also blinded as to the group assignment of the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Biofeedback, Massed->Distributed (Experimental): Sequenced biofeedback Mass Practice--> Distributed Scheduling
  Interventions: Behavioral: Biofeedback; Behavioral: Massed --> Distributed Practice
- No Biofeedback, Distributed (Active Comparator): Speech Motor Chaining with no biofeedback. 2 sessions/wk for 10 weeks
  Interventions: Behavioral: Speech Motor Chaining without Biofeedback; Behavioral: Distributed Practice
- Biofeedback, Distributed (Experimental): Sequenced biofeedback, 2 sessions/wk for 10 weeks
  Interventions: Behavioral: Biofeedback; Behavioral: Distributed Practice
- No Biofeedback, Massed-> Distributed (Experimental): Speech Motor Chaining with no biofeedback. Mass Practice--> Distributed Scheduling
  Interventions: Behavioral: Speech Motor Chaining without Biofeedback; Behavioral: Massed --> Distributed Practice

INTERVENTIONS:
Behavioral: Speech Motor Chaining without Biofeedback — These procedures target sound sequences (consonant-vowel, consonant-consonant, or vowel-consonant). Sessions begin with Pre-practice to elicit the target sounds, with verbal cueing and shaping strategies. The Practice component then includes chaining that is response-contingent. Participants practice in blocks of 6 consecutive trials beginning at the syllable level. If 5/6 are correct, the participant advances to monosyllabic word practice, then multisyllabic word practice, phrase practice, and sentence practice (with the target syllable embedded within each level of complexity). If fewer than 5/6 trials are correct, a different syllable with the target sound pattern is practiced next. Verbal feedback is faded from 5 of 6 trials at the syllable level to only 3 of 6 trials at the sentence level. For more description, see http://speechproductionlab.syr.edu/Resources%20for%20Researchers.html
  Arms: No Biofeedback, Distributed; No Biofeedback, Massed-> Distributed
Behavioral: Biofeedback — Real-time images of the tongue are made available using ultrasound placed beneath the chin. Participants practice speech movements and can be cued to modify their tongue shape or position to achieve clearer speech. Practice structure is similar to the Speech Motor Chaining procedures, but with the addition of a visual reference.
  Arms: Biofeedback, Distributed; Biofeedback, Massed->Distributed
Behavioral: Distributed Practice — 2 sessions per week for 10 weeks
  Arms: Biofeedback, Distributed; No Biofeedback, Distributed
Behavioral: Massed --> Distributed Practice — Week 1: 10 hours of treatment Week 2: 3 hours of treatment Week 3: 3 hours of treatment Week 4: 2 hours of treatment Week 5: 2 hours of treatment
  Arms: Biofeedback, Massed->Distributed; No Biofeedback, Massed-> Distributed

SUMMARY:
The study will test two modifications to speech therapy for 40 school-age children with childhood apraxia of speech to determine how to improve treatment outcomes. The study will compare treatment that includes real-time visual feedback of the tongue during speech using ultrasound vs traditional therapy that does not include ultrasound visual feedback. Additionally, some children will be treated with a traditional schedule of 2 sessions per week, whereas others will be provided with treatment that begins with intensive training (10 hours of therapy in one week) and progresses to a more distributed treatment schedule.

DETAILED DESCRIPTION:
Childhood apraxia of speech is a developmental speech sound disorder that may lead to persisting speech errors, often despite years of treatment. Such impairments may lead to social, academic, and vocational limitations. Thus, there is a need to explore alternate treatment approaches. This study will explore how to improve speech sound production in school-age children with CAS by modifying a standard speech therapy program. Two adaptations to speech therapy will be tested in a 2 x 2 randomized group design.

In Aim 1, a standard treatment schedule of 2 one-hour sessions per week will be compared against a treatment sequence beginning with an intensive therapy schedule (10 hrs of treatment in one week), which will then transition to a more distributed practice schedule. This treatment modification is intended to minimize erred practice between training sessions in the early stages of learning, then foster generalization through increased time between practice sessions.

In Aim 2, a standard treatment that includes only verbal feedback to the client during speech practice will be compared against a treatment sequence that initially includes real-time ultrasound visual feedback of the tongue during speech, which will be faded over the course of treatment. Ultrasound visual feedback is designed to train articulatory movements. It may enhance children's understanding of the articulatory goals of speech movement patterns by comparing executed tongue movements with intended movements. Prior case reports and single subject experimental designs have shown that speech sound production may be enhanced by including ultrasound visual feedback, although no prior randomized group studies have been conducted.

Beside these modifications, the other aspects of treatment will be held constant. Outcomes will be evaluated by tracking changes in percent consonants correct from a large speech sample, scored by individuals who are blind to treatment status. The four groups will be compared to determine the extent to which speech sound therapy can be enhanced through a treatment sequence that begins with intensive practice and/or with ultrasound visual feedback.

ELIGIBILITY:
Inclusion Criteria:

* Native English speakers who hear English as the dominant language in their home setting.
* Must pass a hearing screening.
* Score at or better than -2 standard deviations from the mean on the Matrix Reasoning Task of the Wechsler Abbreviated Scale of Intelligence - 2nd Edition (WASI-2; t-score ≥ 30), Peabody Picture Vocabulary Test - 4th Edition (PPVT-4; standard score ≥ 70), and the Following Directions subtest of the Clinical Evaluation of Language Fundamentals - 5th Edition (CELF-5; scaled score ≥ 3).
* Goldman-Fristoe Test of Articulation - 3rd Edition (GFTA-3) percentile ≤ 5th).
* A diagnosis of CAS will be verified based on a polysyllable picture naming task, diadochokinetic task (puh-tuh-kuh), and syllable repetition task.

Exclusion Criteria:

* Parent report or direct evaluation reveals oral-facial structural abnormalities (e.g., cleft palate).
* Parental report of neurobehavioral disorders (e.g., autism spectrum disorders, ADHD, obsessive-compulsive disorder), or vision problems that are corrected with glasses/contacts.
* Fail a hearing screening, or failure to meet criteria listed above as Inclusionary

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-06-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Syracuse University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Preston JL, Leece MC, Maas E. Intensive Treatment with Ultrasound Visual Feedback for Speech Sound Errors in Childhood Apraxia. Front Hum Neurosci. 2016 Aug 30;10:440. doi: 10.3389/fnhum.2016.00440. eCollection 2016. PMID 27625603
- [Background] Preston JL, Leece MC, McNamara K, Maas E. Variable Practice to Enhance Speech Learning in Ultrasound Biofeedback Treatment for Childhood Apraxia of Speech: A Single Case Experimental Study. Am J Speech Lang Pathol. 2017 Aug 15;26(3):840-852. doi: 10.1044/2017_AJSLP-16-0155. PMID 28715554
- See also: Speech Motor Chaining Procedural manual — http://speechproductionlab.syr.edu/Resources.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Biofeedback, Massed->Distributed, Face-to-Face: Sequenced biofeedback Mass Practice--> Distributed Scheduling
  Biofeedback: Real-time images of the tongue are made available using ultrasound placed beneath the chin. Participants practice speech movements and can be cued to modify their tongue shape or position to achieve clearer speech. Practice structure is similar to the Speech Motor Chaining procedures, but with the addition of a visual reference.
  Massed --> Distributed Practice: Week 1: 10 hours of treatment Week 2: 3 hours of treatment Week 3: 3 hours of treatment Week 4: 2 hours of treatment Week 5: 2 hours of treatment
  Modality: Face-to-Face
- No Biofeedback, Distributed, Face-to-Face: Speech Motor Chaining with no biofeedback. 2 sessions/wk for 10 weeks
  Speech Motor Chaining without Biofeedback: These procedures target sound sequences (consonant-vowel, consonant-consonant, or vowel-consonant). Sessions begin with Pre-practice to elicit the target sounds, with verbal cueing and shaping strategies. The Practice component then includes chaining that is response-contingent. Participants practice in blocks of 6 consecutive trials beginning at the syllable level. If 5/6 are correct, the participant advances to monosyllabic word practice, then multisyllabic word practice, phrase practice, and sentence practice (with the target syllable embedded within each level of complexity). If fewer than 5/6 trials are correct, a different syllable with the target sound pattern is practiced next. Verbal feedback is faded from 5 of 6 trials at the syllable level to only 3 of 6 trials at the sentence level.
  Distributed Practice: 2 sessions per week for 10 weeks
  Modality: Face-to-Face
- Biofeedback, Distributed, Face-to-Face: Sequenced biofeedback, 2 sessions/wk for 10 weeks
  Biofeedback: Real-time images of the tongue are made available using ultrasound placed beneath the chin. Participants practice speech movements and can be cued to modify their tongue shape or position to achieve clearer speech. Practice structure is similar to the Speech Motor Chaining procedures, but with the addition of a visual reference.
  Distributed Practice: 2 sessions per week for 10 weeks
  Modality: Face-to-Face
- No Biofeedback, Massed-> Distributed, Face-to-Face: Speech Motor Chaining with no biofeedback. Mass Practice--> Distributed Scheduling
  Speech Motor Chaining without Biofeedback: These procedures target sound sequences (consonant-vowel, consonant-consonant, or vowel-consonant). Sessions begin with Pre-practice to elicit the target sounds, with verbal cueing and shaping strategies. The Practice component then includes chaining that is response-contingent. Participants practice in blocks of 6 consecutive trials beginning at the syllable level. If 5/6 are correct, the participant advances to monosyllabic word practice, then multisyllabic word practice, phrase practice, and sentence practice (with the target syllable embedded within each level of complexity). If fewer than 5/6 trials are correct, a different syllable with the target sound pattern is practiced next. Verbal feedback is faded from 5 of 6 trials at the syllable level to only 3 of 6 trials at the sentence level. For more description, see http://speechproductionlab.syr.edu/Resources%20for%20Researchers.html
  Massed --> Distributed Practice: Week 1: 10 hours of treatment Week 2: 3 hours of treatment Week 3: 3 hours of treatment Week 4: 2 hours of treatment Week 5: 2 hours of treatment
  Modality: Face-to-Face
- No Biofeeedback, Distributed, Telepractice: Speech Motor Chaining with no biofeedback. 2 sessions/wk for 10 weeks
  Speech Motor Chaining without Biofeedback: These procedures target sound sequences (consonant-vowel, consonant-consonant, or vowel-consonant). Sessions begin with Pre-practice to elicit the target sounds, with verbal cueing and shaping strategies. The Practice component then includes chaining that is response-contingent. Participants practice in blocks of 6 consecutive trials beginning at the syllable level. If 5/6 are correct, the participant advances to monosyllabic word practice, then multisyllabic word practice, phrase practice, and sentence practice (with the target syllable embedded within each level of complexity). If fewer than 5/6 trials are correct, a different syllable with the target sound pattern is practiced next. Verbal feedback is faded from 5 of 6 trials at the syllable level to only 3 of 6 trials at the sentence level.
  Distributed Practice: 2 sessions per week for 10 weeks
  Modality: Telepractice
- No Biofeedback, Massed->Distributed, Telepractice: Speech Motor Chaining with no biofeedback. Mass Practice--> Distributed Scheduling
  Speech Motor Chaining without Biofeedback: These procedures target sound sequences (consonant-vowel, consonant-consonant, or vowel-consonant). Sessions begin with Pre-practice to elicit the target sounds, with verbal cueing and shaping strategies. The Practice component then includes chaining that is response-contingent. Participants practice in blocks of 6 consecutive trials beginning at the syllable level. If 5/6 are correct, the participant advances to monosyllabic word practice, then multisyllabic word practice, phrase practice, and sentence practice (with the target syllable embedded within each level of complexity). If fewer than 5/6 trials are correct, a different syllable with the target sound pattern is practiced next. Verbal feedback is faded from 5 of 6 trials at the syllable level to only 3 of 6 trials at the sentence level. For more description, see http://speechproductionlab.syr.edu/Resources%20for%20Researchers.html
  Massed --> Distributed Practice: Week 1: 10 hours of treatment Week 2: 3 hours of treatment Week 3: 3 hours of treatment Week 4: 2 hours of treatment Week 5: 2 hours of treatment
  Modality: Telepractice
Period: Overall Study
Arm/Group | Biofeedback, Massed->Distributed, Face-to-Face | No Biofeedback, Distributed, Face-to-Face | Biofeedback, Distributed, Face-to-Face | No Biofeedback, Massed-> Distributed, Face-to-Face | No Biofeeedback, Distributed, Telepractice | No Biofeedback, Massed->Distributed, Telepractice
Started | 9 | 9 | 10 | 9 | 10 | 9
Completed | 7 | 7 | 8 | 8 | 9 | 9
Not Completed | 2 | 2 | 2 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biofeedback, Massed->Distributed, Face-to-Face | No Biofeedback, Distributed, Face-to-Face | Biofeedback, Distributed, Face-to-Face | No Biofeedback, Massed-> Distributed, Face-to-Face | No Biofeeedback, Distributed, Telepractice | No Biofeedback, Massed->Distributed, Telepractice | Total
Number analyzed (Participants) | 9 | 9 | 10 | 9 | 10 | 9 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.31 (1.0) | 10.85 (1.7) | 12.2 (2.1) | 10.0 (1.1) | 11.05 (2.4) | 11.16 (2.3) | 10.96 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 3 | 4 | 2 | 17
  Male | 6 | 6 | 8 | 6 | 6 | 7 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 2 | 0 | 0 | 3 | 9
  Not Hispanic or Latino | 6 | 8 | 8 | 9 | 9 | 6 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 9 | 8 | 8 | 7 | 6 | 7 | 45
  More than one race | 0 | 1 | 1 | 2 | 3 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 10 | 9 | 10 | 9 | 56
Speech Sound Accuracy [Mean (Standard Deviation); unit: Percent correct] — The primary outcome measure was percent correct for each participant's target sound-positions in untreated phrase. Participants imitated 20 pre-recorded phrases, each containing the target sound pattern 2 times per stimulus (e.g., for /l/ onset, "leave the location"), resulting in 40 attempts at each sound-position. For each session, 3 transcribers independently transcribed in Phon software (Hedlund & Rose, 2022) and accuracy was averaged across transcribers. Instances where IPA symbols for the Actual transcription differed from the Target transcription was scored as incorrect. Population: Participant withdrew after randomization but before baseline collection of this datapoint
  Percent correct
    number analyzed (Participants) | 9 | 9 | 10 | 8 | 10 | 9 | 55
    (all) | 20.2 (7.3) | 21.2 (12.1) | 17.0 (4.3) | 23.2 (7.4) | 28.9 (8.1) | 35.5 (7.8) | 24.3 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: Speech Sound Accuracy
Description: Percent consonants correct for target sounds: The primary outcome measure was percent correct for each participant's target sound-positions in untreated phrase. Participants imitated 20 pre-recorded phrases, each containing the target sound pattern 2 times per stimulus (e.g., for /l/ onset, "leave the location"), resulting in 40 attempts at each sound-position. For each session, 3 transcribers independently transcribed in Phon software (Hedlund & Rose, 2022) and accuracy was averaged across transcribers. Instances where IPA symbols for the Actual transcription differed from the Target transcription was scored as incorrect.
Time Frame: 10 weeks from the start of treatment
Measure: Mean (Standard Error); unit: Percent correct
Arm/Group | Biofeedback, Massed->Distributed, Face-to-Face | No Biofeedback, Distributed, Face-to-Face | Biofeedback, Distributed, Face-to-Face | No Biofeedback, Massed-> Distributed, Face-to-Face | No Biofeeedback, Distributed, Telepractice | No Biofeedback, Massed->Distributed, Telepractice
Number analyzed (Participants) | 7 | 7 | 8 | 8 | 9 | 9
Percent correct | 54.1 (13.5) | 32.5 (14.1) | 26.8 (10.2) | 42.1 (11.1) | 32.50 (7.0) | 43.0 (7.7)
Statistical Analysis 1: Comparison: Biofeedback, Massed->Distributed, Face-to-Face vs No Biofeedback, Distributed, Face-to-Face vs Biofeedback, Distributed, Face-to-Face vs No Biofeedback, Massed-> Distributed, Face-to-Face vs No Biofeeedback, Distributed, Telepractice vs No Biofeedback, Massed->Distributed, Telepractice; Main effect of biofeedback at 10 weeks; Test type: Superiority; p = .132, Mixed Models Analysis; Mean Difference (Final Values) = -10.0, 95% CI 2-sided [-23.2 to 3.1]
Statistical Analysis 2: Comparison: Biofeedback, Massed->Distributed, Face-to-Face vs No Biofeedback, Distributed, Face-to-Face vs Biofeedback, Distributed, Face-to-Face vs No Biofeedback, Massed-> Distributed, Face-to-Face vs No Biofeeedback, Distributed, Telepractice vs No Biofeedback, Massed->Distributed, Telepractice; Main effect of Practice Distribution at 10 weeks; Test type: Superiority; p = .028, Mixed Models Analysis; Mean Difference (Final Values) = -13.7, 95% CI 2-sided [-25.9 to -1.5]
Statistical Analysis 3: Comparison: No Biofeedback, Distributed, Face-to-Face vs No Biofeedback, Massed-> Distributed, Face-to-Face vs No Biofeeedback, Distributed, Telepractice vs No Biofeedback, Massed->Distributed, Telepractice; Main effect comparing telepractice vs face-to-face treatment; Test type: Superiority; p = .187, Mixed Models Analysis; Mean Difference (Final Values) = -10.0, 95% CI 2-sided [-24.9 to 5.0]
Statistical Analysis 4: Comparison: Biofeedback, Massed->Distributed, Face-to-Face vs No Biofeedback, Distributed, Face-to-Face vs Biofeedback, Distributed, Face-to-Face vs No Biofeedback, Massed-> Distributed, Face-to-Face vs No Biofeeedback, Distributed, Telepractice vs No Biofeedback, Massed->Distributed, Telepractice; Interaction of biofeedback and practice distribution at 10 weeks; Test type: Superiority; p = .125, Mixed Models Analysis; Mean Difference (Final Values) = 20.22, 95% CI 2-sided [-5.8 to 46.3]; η2 =.054

ADVERSE EVENTS:
Time Frame: 5 weeks and 10 weeks after the start of treatment
Arm/Group | Biofeedback, Massed->Distributed, Face-to-Face | No Biofeedback, Distributed, Face-to-Face | Biofeedback, Distributed, Face-to-Face | No Biofeedback, Massed-> Distributed, Face-to-Face | No Biofeeedback, Distributed, Telepractice | No Biofeedback, Massed->Distributed, Telepractice
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/10 | 0/9 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/10 | 0/9 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/10 | 0/9 | 0/10 | 0/9

LIMITATIONS AND CAVEATS:
The interruptions due to the COVID-19 pandemic resulted an imbalance in participants in the Ultrasound vs No Ultrasound conditions, which limits statistical power. Participants were not randomized to telepractice vs face-to-face.

Also, the treatment emphasizes speech sound accuracy. There is not a direct focus on teaching other features such as lexical stress. Other approaches, such as Rapid Syllable Transition Training would be more appropriate to address other elements of speech production.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-04-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT03238677/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/77/NCT03238677/SAP_001.pdf